CLINICAL TRIAL: NCT05568498
Title: Probiotic Treatment for Depression and Associated Mood Disorders in Parkinson's Disease
Acronym: ProD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Silke Cresswell, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H17-01853
Record Dates: First submitted 2022-06-15; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease; Depression
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Ecologic® BARRIER 849 (Maize starch, maltodextrin, vegetable protein, potassium chloride, +/- probiotic bacteria (B. bifidum W23, B. lactis W51, B. lactis W52, L. acidophilus W37, L. brevis W63, L. casei W56, L. salivarius W24, Lc. lactis W19, Lc. lactis W58; ≥ 2,5*10^9 colony forming unit (CFU)/g), magnesium sulphate, manganese sulphate.) sachet, two times daily dosing for a total of 2 grams (viable cell count of 2.5 × 10^9 CFU/gram) per day.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo (maize starch, maltodextrin, vegetable protein, magnesium sulphate, manganese sulphate)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Oral probiotic delivered in powdered form.
  Other Names: Ecologic® BARRIER 849
  Arms: Probiotic
Dietary Supplement: Placebo — Oral placebo delivered in powdered form.
  Arms: Placebo

SUMMARY:
This study evaluates the use of an oral multi-strain probiotic in the treatment of depression in individuals with Parkinson's Disease. Participants will be randomized to either 12-week multi-strain probiotic treatment or placebo with an optional fMRI scan.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a complex condition that carries a high burden of neuropsychiatric comorbidities. About a third of individuals living with Parkinson's disease have one or more depressive disorders, resulting in lower quality of life, greater care dependency, and increased caregiver burden. Gastrointestinal dysfunction is very common in Parkinson's. Constipation is experienced by the vast majority of patients and often manifests years before onset of motor symptoms, symptoms suggestive of irritable bowel syndrome are also commonly found in PD. Increased intestinal permeability has been demonstrated in PD. Impaired intestinal barrier function can lead to chronic systemic low-grade inflammation, which has been strongly associated with mood disorders. Several lines of evidence suggest a link between the gut microbiome and Parkinson's disease.

The microbiome has been linked to depression both in human and animal studies. Several studies have found beneficial effects of probiotics on mood disorders in non-PD populations, including stress and depressive behaviour in animal models, and sad mood reactivity and major depressive disorder in humans.

In summary, given the high rate of depression in PD, the growing evidence that probiotics may improve depression and mood disorders in non-PD populations, and the strong links between the gut microbiome and PD, we will carry out a randomized, blinded, placebo-controlled study into the use of a multi-strain probiotic to improve depression and Parkinson's disease.

Recruitment: Approximately 60 participants will be randomized to either the probiotic intervention arm or placebo treatment. Participants will mainly be recruited from the Pacific Parkinson's Research Centre movement disorder clinic at the University of British Columbia in Vancouver.

Participants will receive a detailed description of the study and will need to provide informed consent for participation in the study. Participants will be screened for inclusion and exclusion criteria.

Assessments: Clinical assessments of motor function, cognition and neuropsychiatric symptoms will be done before the 12 week intervention phase as well as following after the 12 week intervention with regular check ins during the course of the intervention. Blood samples and stool samples will be collected before and after the intervention. An optional fMRI scan will be completed at the first and last study visit, pre- and post-intervention.

The primary outcome will be the difference between the probiotic vs. placebo groups in mean Inventory of Depressive Symptomatology - Clinician-Rated (IDS-C) pre-/post-intervention. The primary analysis will be based on intention-to-treat. For other secondary outcomes, the between-group difference analysis will be applied to the fatigue, anxiety, PD motor function, severity (UPDRS I-III) and quality of life scores pre/post intervention, respectively. Adverse events, tolerability and drop-out rates will be registered and overall rates compared between the intervention groups. Furthermore, differences and changes in blood markers and microbiome composition will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Parkinson's disease based on UK Brain Bank criteria
2. Between the ages of 40-80 years
3. Hoehn and Yahr stage between 1-3 (mild to moderate PD) in the "ON" state
4. Mild to moderate depression (clinical diagnosis of mild to moderate depression in the MINI clinical interview and/or BDI-II score of 14-28, and/or IDS-C score of 12-36, and/or QIDS-SR score of 6-15 in the "ON" state)
5. Women of childbearing potential must agree to use a medically approved method of birth control (e.g., hormonal contraceptives, intrauterine devices, vasectomy/tubal litigation, barrier methods and double barrier method) and must have negative pregnancy test results at screening and baseline
6. Willingness to maintain current physical activity levels during study period
7. English proficiency

Exclusion Criteria:

1. Atypical parkinsonism
2. Active suicidality
3. Active psychosis
4. Cognitive score (MoCA) of < 21 in the "ON" state
5. Severe depression (BDI-II score > 28 and/or IDS-C score > 36, and/or QIDS-SR score > 15 in the "ON" state)
6. Probiotic, saccharomyces boulardii and/or antibiotic use in the past 3 months (yogurt, kefir, and other probiotic containing foods are allowed)
7. The use of natural health products that affect depression (e.g., St. John's Wort, passion flower, gaba, 5-htp, kava, bacopa, efa's)
8. Change in schedule of concurrent psychotherapy or brain stimulation for the treatment of mood or anxiety disorders in the last 4 weeks
9. Change in antidepressant or anxiolytic medication (including benzodiazepines) within the last 4 weeks
10. Change in Parkinson's medication within the last 2 weeks
11. Neurological disease other than PD, including Alzheimer's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, a brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
12. A significant immune-compromised condition due to either a health condition or use of an immune suppressant (e.g., AIDS, lymphoma, chemotherapy treatment, patients undergoing long-term systemic corticosteroid or immunosuppressant treatment)
13. A known bleeding disorder
14. Current illness (e.g., a cold or flu-like symptoms) and infections (e.g., hepatitis, HIV, gastroenteritis, fungal, or parasitic infections)
15. Allergy to corn starch or corn
16. Concurrent treatment for Parkinson's disease with Duodopa
17. Change in Deep Brain Stimulation (DBS) stimulation parameters in the last 4 weeks
18. New onset of significant psychiatric symptoms following DBS procedure that are considered likely related
19. Women who are pregnant, breast feeding, or planning to become pregnant during the course of the trial
20. Unstable medical conditions or serious disease/conditions (e.g., cancer undergoing active treatment, poorly controlled diabetes)
21. Drug and/or substance abuse
22. Claustrophobia inhibiting ability to complete an MRI
23. The patient, in the opinion of the Investigator, is unable to adhere to the requirements of the study. This includes any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a significant language barrier or cognitive impairment

4.2.1 Additional Exclusion Criteria for Magnetic Resonance Imaging (MRI)

The criteria below will also be reviewed with the MRI technologist before any scanning can occur.

Absolute Contraindications:

1. Cardiac pacemaker, wires, or defibrillator
2. Metal in eye or orbit
3. Ferromagnetic aneurysm clip
4. Pregnancy
5. Makeup tattoos that are not designed to fade over time
6. Copper or stainless steel intrauterine device

Relative Contraindications (participation depends on the individual situation):

1. Artificial heart valve
2. Ear or eye implant
3. Brain aneurysm clip
4. Implanted electronic device (e.g., drug infusion pump, electrical stimulator)
5. Coil, catheter, or filter in any blood vessel
6. Orthopedic hardware (artificial joint, plate, screw, rod)
7. Shrapnel, bullets, or other metal fragments
8. Surgery, medical procedure, or tattoos (including tattooed eyeliner) in the last six weeks
9. Other metallic prostheses

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology - Clinician-Rated (IDS-C) | 13 weeks
  The Inventory for Depressive Symptomatology is a measure of depressive signs and symptoms administered by a trained clinician. The Score range is 0-84 points with a higher score indicating greater levels of depressive symptomatology.

SECONDARY OUTCOMES:
Beck Depression Inventory, 2nd Edition (BDI-II) | 13 weeks
  The Beck Depression Inventory is a self-reported 21-question multiple-choice self-report inventory on a scale from 0-63. A higher score indicates greater characteristic attitudes and symptoms of depression.
Fatigue Severity Scale (FSS) | 13 weeks
  The Fatigue Severity Scale is a self-reported 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders on a scale from 1 (strongly disagree) to 7 (strongly agree). The minimum score is 9 and the maximum score is 63. A higher score indicates greater fatigue severity.
Montreal Cognitive Assessment (MoCA) | 13 weeks
  The Montreal Cognitive Assessment test is a one-page 30-point assessment administered by trained individuals that is used for detecting cognitive impairment. Score may range from 0-30 points and a lower score may indicate greater cognitive impairment.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 13 weeks
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale is a clinical assessment of motor and non-motor symptoms in individuals with Parkinson's Disease. It consists of four subscales. Subscales 1, 3, and 4 are administered by a trained individual and subscale 2 is self-reported. Each item is rated from 0 to 4. Total score can range from 0-199 with a higher score indicating greater impairment in Parkinson's disease.
Parkinson's Anxiety Scale (PAS) | 13 weeks
  The Parkinson's Anxiety Scale is a 12-point observer or patient-rated scale that has three subscales: persistent anxiety, episodic anxiety, and avoidance behavior; It is rated using a Likert scale (0-4). Possible scores range from 0-48 with a higher score indicating greater severity of anxiety symptoms.
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 13 weeks
  The Parkinson's Disease Quality of Life Questionnaire is a self-reported questionnaire that assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. It consists of 39 items which are rated on a Likert scale (0-4). Each dimension's score can range from 0-100. Higher score indicates worse quality of life.

IPD SHARING:
Plan to Share IPD: No